CLINICAL TRIAL: NCT05417139
Title: Sintilimab Combined With Chemotherapy and Radiotherapy in Newly Diagnosed Metastatic Nasopharyngeal Carcinoma: A Multicenter Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); First People's Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Fang-Yun Xie, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2021-382
Record Dates: First submitted 2022-06-07; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immunotherapy+induction chemotherapy+radiotherapy (Experimental)
  Interventions: Other: Immunotherapy+induction chemotherapy+radiotherapy

INTERVENTIONS:
Other: Immunotherapy+induction chemotherapy+radiotherapy — All enrolled patients received Sintilimab (200mg, d1, q3w) + GP (gemcitabine 1000mg / m2, d1, d8 + cisplatin 80mg / m2, d1, q3w) for 4-6 cycles followed by radiotherapy of primary site and cervical metastasis, and Sintilimab (200mg, q3w) treatment was continued during and after radiotherapy until disease progression or toxicity or up to 2 years.

SUMMARY:
To explore the progression-free survival rate (progression-free survival, PFS), overall survival (OS), objective response rate(objective response rate, ORR) and safety of patients with Sintilimab + GP chemotherapy combined with radiotherapy for newly diagnosed metastatic NPC.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically diagnosed nasopharyngeal cancer with distant metastasis; not received anticancer treatment.
* ECOG Score (PS score) 0 or 1.
* Neutrophil count > 1.5*10^9/L, hemoglobin > 90g/L, and platelet count > 100*10^9/L.
* ALT or AST level < 2.5 times upper normal limit (upper limit of normal, ULN), bilirubin level < 1.5 times ULN.
* Creatinine clearance level > 60 ml/min.
* Patients must sign an informed consent and must be willing and able to comply with the visit, treatment protocol, laboratory tests and other requirements specified in the study protocol.
* Pregnant female subjects must agree to use reliable contraception within 1 year from the screening visit to the last Sintilimab administration.

Exclusion Criteria:

* Age> 65 years old or <18 years old.
* HBsAg positive and HBV DNA> 10*10^3 copy number/ml.
* HCV antibody positive.
* Active, known, or suspected autoimmune diseases. Subjects with type I diabetes, hypothyroidism with only hormone replacement therapy, and skin disease without systemic treatment (such as vitiligo, psoriasis, or alopecia) can be selected.
* A history of interstitial lung disease.
* Received systemic hormone or other immunosuppressive therapy with an equivalent dose of> 10mg of prednisone per day within 28 days prior to signing the informed consent. Subjects with a systemic hormone dose of 10mg prednisone per day or inhaled / topical corticosteroids may be enrolled.
* Received or will be vaccinated within 30 days before signing the informed consent.
* Pregnancy or breastfeeding women (pregnancy tests should be considered).
* Other malignancies within 5 years, except carcinoma in situ, fully treated non-melanoma skin cancer, and papillary thyroid carcinoma.
* previous allergies to macromolecular protein preparations, or any component of Sintilimab.
* Human immunodeficiency virus (HIV) infection.
* Other conditions that may affect the safety or trial compliance of the subject, including symptomatic heart failure, unstable angina, myocardial infarction, active infection requiring systemic treatment, mental illness or family and social factors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 1-year PFS
  from enrollment of treatment to the first disease progression, death, or the last follow-up

SECONDARY OUTCOMES:
OS | 1-year OS
  from enrollment treatment to death of any cause, if not, to last follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China